CLINICAL TRIAL: NCT00478309
Title: Gene Environment Risk Assessment and CRC Screening
Brief Title: Genetic Epidemiology Risk Assessment Program or Usual Care in Colorectal Cancer Screening for Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000538405; IRB#06807 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Cancer; Healthy, no Evidence of Disease
Keywords: colon cancer; rectal cancer; healthy, no evidence of disease
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Counseling; Early Intervention, Educational

ARMS (2):
- Arm I (No Intervention): Participants receive standard primary care.
- Arm II (Experimental): Participants receive standard primary care followed by the Genetic Epidemiology and Risk Assessment (GERA) intervention. Participants also participate in a discussion session regarding the GERA including the rationale behind methylenetetrahydrofolate reductase mutation detection and folate assessment and its relationship to colorectal cancer risk.
  Interventions: Other: counseling intervention; Other: educational intervention

INTERVENTIONS:
Other: counseling intervention
  Arms: Arm II
Other: educational intervention
  Arms: Arm II

SUMMARY:
RATIONALE: The Genetic Epidemiology and Risk Assessment program may be more effective than usual care in increasing the number of healthy participants who regularly receive screening for colorectal cancer.

PURPOSE: This randomized clinical trial is studying the Genetic Epidemiology and Risk Assessment program to see how well it works compared with usual care to increase colorectal cancer screening in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare Genetic Epidemiology and Risk Assessment (GERA) feedback vs usual care (UC) in terms of colorectal cancer (CRC) screening utilization by healthy participants.
* Determine the impact of GERA feedback and UC on psychological distress in these participants.
* Compare GERA feedback vs UC in terms of intention to have CRC screening, perceived CRC risk, CRC knowledge, salience and coherence of CRC screening, and support for CRC screening in these participants.
* Identify factors that moderate the impact of GERA feedback on CRC screening utilization.

OUTLINE: This is a randomized study. Participants are randomized to 1 of 2 screening arms.

* Arm I: Participants receive standard primary care.
* Arm II: Participants receive standard primary care followed by the Genetic Epidemiology and Risk Assessment (GERA) intervention. Participants also participate in a discussion session regarding the GERA including the rationale behind methylenetetrahydrofolate reductase mutation detection and folate assessment and its relationship to colorectal cancer risk.

All participants undergo a fecal occult blood test 3 weeks after the screening office visit.

PROJECTED ACCRUAL: A total of 1,950 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participants meeting the following criteria:

  * No personal history of colorectal polyps or cancer or inflammatory bowel disease
  * No family history of familial adenomatous polyposis, hereditary nonpolyposis colorectal cancer (CRC), or CRC in more than 1 first-degree relative
* Nonadherent with standard CRC screening recommendations at the time of their index office visit

PATIENT CHARACTERISTICS:

* Able to communicate with ease in English

PRIOR CONCURRENT THERAPY:

* More than 6 weeks since prior antibiotics or antifolate medications (e.g., sulfasalazine, methotrexate)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 697 (Actual)
Dates: Start 2007-03; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Comparison of Genetic Epidemiology and Risk Assessment (GERA) feedback vs usual care (UC) in terms of colorectal cancer (CRC) screening utilization | At study completion
Impact of GERA feedback and UC on psychological distress | At study completion
Comparison of GERA feedback vs UC in terms of intention to have CRC screening, perceived CRC risk, CRC knowledge, salience and coherence of CRC screening, and support for CRC screening | At study completion
Factors that moderate the impact of GERA feedback on CRC screening utilization | At study completion

CONTACTS AND LOCATIONS:
Overall Officials: David Weinberg, MD, MSC, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Myers RE, Manne SL, Wilfond B, Sifri R, Ziring B, Wolf TA, Cocroft J, Ueland A, Petrich A, Swan H, DiCarlo M, Weinberg DS. A randomized trial of genetic and environmental risk assessment (GERA) for colorectal cancer risk in primary care: trial design and baseline findings. Contemp Clin Trials. 2011 Jan;32(1):25-31. doi: 10.1016/j.cct.2010.08.013. Epub 2010 Sep 7. PMID 20828635